CLINICAL TRIAL: NCT06894121
Title: Comparison of the Efficacy of Unilateral and Bilateral Proximal Greater Occipital Nerve Pulsed Radiofrequency in the Treatment of Migraine
Brief Title: Comparing Unilateral and Bilateral Proximal GONPRF in Migraine Treatment
Acronym: (UBGON-PRF)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ülkü Sabuncu, Assoc. Prof. Dr., Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TABED 1-24-763
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-12

CONDITIONS: Migraine, Greater Occipital Nerve Pulsed Radiofrequency; Headache Disorders; Ultrasound Guided Nerve Block
Keywords: GON PRF; Migraine Treatment; Headache Pain Management; Ultrasound-Guided GON Pulsed Radiofrequency
MeSH Terms: conditions — Migraine Disorders; Headache Disorders

STUDY DESIGN:
Intervention Model Description: This study will have two arms comparing the efficacy of unilateral GON PRF treatment with bilateral GON PRF treatment. The clinical outcomes of the treatment methods in each arm will be evaluated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unilateral GON PRF Treatment (Other): This arm involves applying unilateral greater occipital nerve pulsed radiofrequency (GON PRF) at the C2 level using ultrasound guidance. The procedure is performed on one side of the head (unilateral).
  Interventions: Other: Greater Occipital Nerve Pulsed Radiofrequency (Unilateral)
- Bilateral GON PRF Treatment (Experimental): This arm involves applying bilateral greater occipital nerve pulsed radiofrequency (GON PRF) at the C2 level using ultrasound guidance. The procedure is performed on both sides of the head (bilateral).
  Interventions: Other: Bilateral GON PRF Treatment:

INTERVENTIONS:
Other: Greater Occipital Nerve Pulsed Radiofrequency (Unilateral) — Greater Occipital Nerve (GON) Pulsed Radiofrequency (PRF) treatment is performed under sterile conditions in the operating room. The patient is positioned in the prone position with neck flexion. Under ultrasound guidance at the proximal (C2) level, the needle is carefully placed near the GON, targeting the space between the Obliquus Capitis Inferior (OCI) muscle and C2's bifid spinous process. After proper sterilization, a linear ultrasound probe is used transversely over the occipital protuberance to locate the C1 and C2 vertebrae. Once identified, the RF needle and electrode are inserted laterally to medially using in-plane technique. A sensory stimulation test is done, and the PRF therapy is applied at a 45V setting, 5 Hz, and 5 ms pulse width for 360 seconds, with a maximum temperature of 42°C. No drug injections are administered during the procedure. Post-procedure, the patient is monitored for at least 1 hour before discharge after a general and neurological evaluation.
  Other Names: UGON-PRF
  Arms: Unilateral GON PRF Treatment
Other: Bilateral GON PRF Treatment: — Greater Occipital Nerve (GON) Pulsed Radiofrequency (PRF) treatment is performed under sterile conditions in the operating room. The patient is positioned in the prone position with neck flexion. Under ultrasound guidance at the proximal (C2) level, the needle is carefully placed near the GON, targeting the space between the Obliquus Capitis Inferior (OCI) muscle and C2's bifid spinous process. After proper sterilization, a linear ultrasound probe is used transversely over the occipital protuberance to locate the C1 and C2 vertebrae. Once identified, the RF needle and electrode are inserted laterally to medially using in-plane technique. A sensory stimulation test is done, and the PRF therapy is applied at a 45V setting, 5 Hz, and 5 ms pulse width for 360 seconds, with a maximum temperature of 42°C. No drug injections are administered during the procedure. Post-procedure, the patient is monitored for at least 1 hour before discharge after a general and neurological evaluation.
  Bilater
  Other Names: BGON-PRF
  Arms: Bilateral GON PRF Treatment

SUMMARY:
This study is designed to compare the clinical effectiveness of unilateral and bilateral Greater Occipital Nerve Pulsed Radiofrequency (GON-PRF) treatment at the C2 level in patients with migraine. The procedure will be guided by ultrasound and will focus on evaluating how each technique affects migraine symptoms.

The main goal of this study is to assess the impact of both unilateral and bilateral GON-PRF treatments on migraine relief. Additionally, the secondary objectives of this study include evaluating the effects of these treatments on migraine-related disability and comparing any potential side effects or complications that may occur during the treatments.

This research will help us understand which technique may be more effective and provide more information on the safety of these treatments.

DETAILED DESCRIPTION:
Migraine is a common neurological disorder that can affect patients' quality of life and socio-economic functionality. In cases of resistant headaches that do not respond to conservative pharmacological treatment, peripheral nerve blocks, particularly greater occipital nerve (GON) block, can be applied. GON block (GONB) can help reduce the frequency and intensity of attacks, as well as the systemic side effects of pharmacological treatment. However, the literature reports that the effectiveness of GON block with local anesthetics and steroids for the treatment of various headache disorders is limited to a few weeks to several months .

To prolong the effect of peripheral nerve blocks, pulsed radiofrequency (PRF) is used. PRF modulates pain transmission without damaging the nerve or surrounding sensitive structures by creating an electrical field in the targeted nerves. Greater occipital nerve pulsed radiofrequency (GON PRF) has been found to be effective and safe in the treatment of migraine . In the treatment of migraine resistant to conservative treatment, GON block and GON PRF, both proven to be effective and safe, are widely used in pain management practice and in our clinic.

GON block and GON PRF can be performed using anatomical landmark technique or under ultrasound guidance (USG). Currently, two different techniques for ultrasound-guided GON block are described. These are the proximal technique targeting the GON at the second cervical vertebra (C2) level and the distal technique targeting the superior nuchal line level. It has been reported that GON block and GON PRF applied with the proximal technique under ultrasound guidance are effective. In our clinic, we apply GON block and GON PRF treatments using ultrasound guidance with either the proximal or distal technique.

Although the exact mechanism of long-term headache relief following peripheral nerve blocks is unknown, it is thought to be related to central pain modulation. The upper cervical nerve roots are anatomically and functionally connected to the trigeminal pathways, and they converge in the trigeminal cervical complex. In a neurophysiological study conducted by Busch et al. on fifteen healthy volunteers without headaches, it was found that unilateral nerve block causes bilateral inhibition, and this inhibitory effect is thought to be due to modulation of the heterosynaptic convergence transmission of second-order neurons or interneurons extending from the caudal trigeminal nucleus to the upper cervical segments. In a retrospective study conducted on chronic migraine patients, it was reported that unilateral GONB was as effective as bilateral GONB in terms of the frequency, severity, and duration of headaches, with the added benefit of a lower frequency of side effects with unilateral GONB. Another retrospective study compared unilateral and bilateral proximal GON block in the treatment of chronic migraine. It was found that proximal GON block at the C2 level was effective in the treatment of chronic migraine, and bilateral application was not superior to unilateral application, with patients tolerating unilateral blocks better.

In our clinic, GON PRF treatment is performed under sterile conditions in an operating room, with patients monitored during the procedure and intravenous access established. For the proximal (C2) level, patients are positioned in a prone position with neck flexion. Anatomical landmarks include the obliquus capitis inferior (OCI) muscle and the bifid spinous process of C2. After sterilizing the application area, a linear ultrasound probe is placed transversely on the occipital protuberance, and it is moved caudally in the sagittal plane to first visualize C1 with a single spinous process, and then, when moving further caudally, C2 with two spinous processes. The probe is then moved laterally to visualize the OCI and semispinalis capitis (SSC) muscles, and it is slightly directed cephalad. The GON appears as an oval, hypoechoic structure between the OCI and SSC muscles at this level and is selected as the target. A catheter needle (22 gauge 5 cm 5 mm active tip RF cannula) and RF electrode are placed using an in-plane technique, from lateral to medial, near the target area (right or left GON). Following this, a sensory stimulation test is performed using the RF generator. After reporting dysesthesia and tingling sensations in the occipital region below 0.2 V by the patient, PRF treatment is applied at 45 V, 5 Hz, and 5 ms pulse width for 360 seconds, ensuring that the electrode tips do not exceed 42°C. For bilateral GON PRF, the same procedure is applied to the other side. No drug injections are administered during the GON PRF treatment. After the procedure, patients are observed in the recovery room for at least one hour and are discharged following a general and neurological evaluation.

According to current knowledge, there is no study comparing the effectiveness of unilateral and bilateral GON PRF in the treatment of migraine. Therefore, our study primarily aims to prospectively compare the clinical efficacy of unilateral and bilateral GON PRF treatment performed at the C2 level using a proximal technique under ultrasound guidance in migraine patients. Additionally, secondary objectives of this study include evaluating the effects of unilateral and bilateral GON PRF treatments on migraine-related disability and comparing any potential side effects and complications associated with the treatment.

ELIGIBILITY:
Inclusion Criteria:Volunteers who are followed up at the Algology polyclinic of Ankara Bilkent City Hospital, between the ages of 18-65, who meet the diagnosis criteria for episodic (≥5 attacks/month) or chronic migraine according to ICHD-3 criteria, who do not benefit sufficiently from the migraine prevention medications used, who are not currently using migraine prevention medications or who have not changed their medication and/or dosage in the last 3 months, who do not have bleeding-clotting disorders and active infection in laboratory tests, who are not pregnant or suspected of being pregnant, who do not have a history of craniocervical surgery that may disrupt the anatomical structure in the intervention area, who can understand and approve the treatment and the informed consent form and who can comply with the treatment will be included in this study. Exclusion criteria for files/records/materials to be included in the study: Patients with a history of primary headache other than migraine according to ICHD-3 criteria, <5 attacks per month, comorbid diseases that may cause headaches (such as uncontrolled hypertension, intracranial lesions), and those who have received interventional treatment, botulinum toxin injection and/or non-pharmacological treatment (acupuncture, physical therapy, ozone, cognitive behavioral therapy, etc.) for migraine within 3 months prior to GON-PRF treatment will not be included in the study.

-

Exclusion Criteria:The voluntary participants' request to withdraw for any reason at any stage of the study, the volunteer/legal representative's withdrawal of consent to participate in the study, failure to attend follow-up, and the emergence of any of the following criteria for not being included in the study.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | Baseline, 3 months.
  The Visual Analog Scale (VAS) is used to assess the severity of migraine pain in patients, with scores ranging from 0 to 10. A score of 0 represents no pain, while a score of 10 represents the worst pain imaginable. This scale is used to monitor changes in pain intensity before and after treatment

SECONDARY OUTCOMES:
The Migraine Disability Assessment Scale (MIDAS) | Baseline, 3 months.
  The Migraine Disability Assessment Scale (MIDAS) is designed to evaluate the impact of migraines on a patient's ability to perform daily activities. It quantifies disability based on the frequency and severity of migraines over a specific period. This scale helps to assess how migraines interfere with a patient's work, social, and household activities

CONTACTS AND LOCATIONS:
Overall Officials: Sukriye Dadali, M.D., Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Health Sciences University, Ankara Bilkent City Hospital, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers due to confidentiality constraints and data protection policies.

REFERENCES:
- [Background] Oliveira K, Dhondt N, Englesakis M, Goel A, Hoydonckx Y. Pulsed Radiofrequency Neuromodulation of the Greater Occipital Nerve for the Treatment of Headache Disorders in Adults: A Systematic Review. Can J Pain. 2024 May 15;8(1):2355571. doi: 10.1080/24740527.2024.2355571. eCollection 2024. PMID 38915302